CLINICAL TRIAL: NCT01932073
Title: Low-Level Laser Therapy for the Management of Radiation Dermatitis: A Pilot Study in Breast Cancer Patients
Brief Title: Laser Therapy for the Management of Radiation Dermatitis
Acronym: DERMIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Prof. dr. Jeroen Mebis, MD, PhD, Hasselt University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13.43/onco13.05
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Radiation Dermatitis
Keywords: Radiation; dermatitis; radiodermatitis; radiotherapy induced; skin reactions; low level laser therapy; breast cancer
MeSH Terms: conditions — Radiodermatitis; Dermatitis; Breast Neoplasms | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Receives institutional skin care protocol
- Treatment Group (Experimental): Receives institutional skin care protocol and, when applicable (if skin reactions develop), Low-Level Laser Therapy
  Interventions: Device: Low-Level Laser Therapy

INTERVENTIONS:
Device: Low-Level Laser Therapy — Low-Level Laser Therapy will be applied, twice a week, from the moment skin reactions become painful until skin reactions are no longer painful
  Arms: Treatment Group

SUMMARY:
Low Level Laser Therapy (LLLT) is a form of phototherapy which involves the application of light to injuries and lesions to promote tissue regeneration. It is a noninvasive treatment modality based on the photochemical effect of light on tissues, which modulates various metabolic processes.

LLLT has been used for a wide range of conditions, in particular in dermatology, to promote wound healing, reduce inflammation and oedema, and relieve pain. In this study, we intend to assess the efficacy of LLLT to manage radiotherapy-induced skin reactions (or radiation dermatitis), a very common and distressing side effect of cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of noninvasive (Stage 0) or invasive (Stages 1, 2 or 3A) breast adenocarcinoma
* Treatment with primary breast-sparing surgery (lumpectomy) and/ or neoadjuvant (preoperative) or adjuvant (postoperative) chemotherapy or hormonal treatment
* Scheduled for postoperative radiotherapy with standard technique (isocentric) and fractionation regime (i.e., 25 daily fractions to the whole breast followed by a boost of 8 fractions to the tumor bed, 2 Gy per fraction, five times per week)
* Provide signed informed consent

Exclusion Criteria:

* Previous irradiation to the same breast
* Metastatic disease
* Mastectomy surgery
* Concurrent chemo-radiotherapy
* Required use of bolus material to deliver radiation therapy (i.e., material placed on the to-be-irradiated zone to modulate the delivered dose in order to ensure an optimal distribution of the radiation dose)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2013-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Radiation Dermatitis Grade | 3 months (during radiation therapy and one month after)
  objective scoring of the severity of radiation dermatitis using the grading system of the Radiation Therapy Oncology Group/ European Organization for Research and Treatment of Cancer (RTOG/ EORTC).
Radiation Dermatitis Assessment | 3 months (during radiation therapy and one month after)
  Radiation dermatitis assessment scale (Radiation-Induced Skin Reaction Assessment Scale, RISRAS)
Pain | 3 months (during radiation therapy and one month after)
  evaluation of pain using a visual analogue scale

SECONDARY OUTCOMES:
Quality of Life | 3 months (during radiation therapy and one month after)
  Health-related quality of life measure specific to skin diseases (Skindex-16)
Impact of Radiation Dermatitis | 3 months (during radiation therapy and one month after)
  Self-report on the impact of radiation dermatitis on daily activities
Satisfaction with therapy | 3 months (during radiation therapy and one month after)
  Self-report on the efficacy of and the global satisfaction with the management of radiation dermatitis

OTHER OUTCOMES:
Moist desquamation | 6.5 weeks (during radiation therapy)
  Onset time of moist desquamation

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Mebis, MD, PhD, Principal Investigator — Jessa Hospital
Locations (1):
- Jessa Hospital - Oncology department, Hasselt, Belgium